CLINICAL TRIAL: NCT03255512
Title: Multi-center, Randomized, Placebo-controlled, Double-blind Group Comparison Study to Investigate Safety, Tolerability and Blood Pressure of 2.5 mg, 5.0 mg and 10 mg Vericiguat Each Given Over 14 ± 3 Days Together With Isosorbite Mononitrate (ISMN) 60 mg Extended Release Formulation After a Pretreatment Phase (ISMN-starting Dose: 30 mg) in Stable Coronary Artery Disease (CAD) Patients With or Without Heart Failure Aged 30 to 80 Years - Vericiguat ISOsoRbite Mononitrate Interaction (VISOR) Study
Brief Title: Vericiguat Drug-drug Interaction Study With Isosorbite Mononitrate in Stable Coronary Artery Disease Patients
Acronym: VISOR
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 18582; 2016-005178-36 (EudraCT Number)
Record Dates: First submitted 2017-08-03; First posted 2017-08-21 (Actual); Last update posted 2021-12-29 (Actual); Status verified 2021-12

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease | interventions — vericiguat; isosorbide-5-mononitrate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vericiguat + isosorbite mononitrate (Experimental): Subjects received Isosorbide mononitrate (ISMN) up-titration with 30 mg / 60 mg, about 7 days each,prior to start of vericiguat administration.
  Then subjects received 2.5 mg vericiguat for about 14 days, followed by 5 mg vericiguat for about 14 days, followed by 10 mg vericiguat for about 14 days together 60 mg ISMN od on each day of vericiguat administration, taken 1 hour prior to vericiguat (in-house days) or together with vericiguat (out-patient days).
  Interventions: Drug: Vericiguat (BAY1021189); Drug: Isosorbide mononitrate (ISMN)
- Placebo + isosorbite mononitrate (Placebo Comparator): Subjects received Isosorbide mononitrate (ISMN) up-titration with 30 mg / 60 mg, about 7 days each, prior to start of placebo administration.
  Then subjects received placebo matching 2.5 mg vericiguat for about 14 days, followed by placebo matching 5 mg vericiguat for about 14 days, followed by placebo matching 10 mg vericiguat for about 14 days together 60 mg ISMN od on each day of placebo administration, taken 1 hour prior to placebo (in-house days) or together with placebo (out-patient days).
  Interventions: Drug: Placebo; Drug: Isosorbide mononitrate (ISMN)

INTERVENTIONS:
Drug: Vericiguat (BAY1021189) — 2.5 mg/tablet; 5 mg/tablet or 10 mg/tablet
  Arms: Vericiguat + isosorbite mononitrate
Drug: Placebo — Matching placebo
  Arms: Placebo + isosorbite mononitrate
Drug: Isosorbide mononitrate (ISMN) — 30 mg/tablet or 60 mg/tablet

SUMMARY:
This study is intended to investigate the pharmacodynamic drug-drug interaction as well as the safety and tolerability of isosorbite mononitrate and vericiguat in patients with stable coronary artery disease.

ELIGIBILITY:
Inclusion Criteria:

Patients with stable CAD defined by

* coronary artery stenosis in any of the 3 main coronary vessels > 50% documented by coronary angiography within last 36 months
* or history of myocardial infarction
* Age: 30 to 80 years (inclusive) at the first screening examination
* Body mass index (BMI): above/equal 18.0 and below/equal 36.0 kg / m²

Exclusion Criteria:

* Intervention e.g. revascularization by percutaneous coronary intervention (PCI) and/or coronary artery bypass graft (CABG) during the last 3 months
* Progressive angina with symptoms of worsening of angina within the < 3 months prior to the first screening examination
* History of recent (< 6 months prior to the first screening examination) myocardial infarction or unstable angina
* Symptomatic carotid stenosis, or transient ischemic attack or stroke within 3 months prior to the first screening examination or patients with stroke at more than 3 months prior to the first screening examination with significant residual neurologic involvement
* Insulin dependent diabetes mellitus
* Clinically relevant cardiac ischemia at screening
* Clinical significant persistent ischemia, which should be ruled out by clinical judgment of the investigator, based on medical history, available clinical data e.g. past angiograms or preexisting or current exercise testing with any imaging technique (e.g. dobutamine stress echocardiography, adenosine or dobutamine stress cardiac magnetic resonance imaging (CMR), scinthigraphy or exercise ECG)
* Atrial fibrillation, pacemaker, defibrillator, atrial ventricular (AV)-block II and III
* Systolic blood pressure below 110 or above 160 mmHg at first screening visit
* Diastolic blood pressure above 100 mmHg at first screening visit
* Heart rate below 50 or above 100 beats / min (taken from ECG measurement) at first screening visit
* Estimated glomerular filtration rate (eGFR) < 30 mL/min/1.73m*2 at first screening visit

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2017-08-17 (Actual); Primary Completion 2018-02-07 (Actual); Study Completion 2018-03-23 (Actual)

PRIMARY OUTCOMES:
Blood pressure | Up to 8 weeks
  Regular measurements of blood pressure after a vericiguat administration on the first and on the last days of each dose step of vericiguat, and on the first days of ISMN up-titration.
Heart rate | Up to 8 weeks
  Regular measurements heart rate after a vericiguat administration on the first and on the last days of each dose step of vericiguat, and on the first days of ISMN up-titration.

SECONDARY OUTCOMES:
Number of participants with adverse events | Up to 9 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (6):
- Germany (6):
  - Universitätsherzzentrum Freiburg - Bad Krozingen, Bad Krozingen, Baden-Wurttemberg
  - Universitätsklinikum Heidelberg, Heidelberg, Baden-Wurttemberg
  - Medizinische Einrichtungen der Universität Bonn, Bonn, North Rhine-Westphalia
  - SocraTec R&D GmbH, Erfurt, Thuringia
  - Charité - Campus Virchow-Klinikum (CVK), Berlin
  - Universitätsklinikum Hamburg Eppendorf (UKE), Hamburg

REFERENCES:
- [Derived] Boettcher M, Mikus G, Trenk D, Dungen HD, Donath F, Werner N, Karakas M, Besche N, Schulz-Burck D, Gerrits M, Hung J, Becker C. Vericiguat in combination with isosorbide mononitrate in patients with chronic coronary syndromes: The randomized, phase Ib, VISOR study. Clin Transl Sci. 2022 May;15(5):1204-1214. doi: 10.1111/cts.13238. Epub 2022 Mar 17. PMID 35299288
- See also: Click here to find results for studies related to Bayer products. — http://clinicaltrials.bayer.com/